CLINICAL TRIAL: NCT06365788
Title: A Multicenter Single Arm Phase II Study With Bicalutamide in Combination With Abemaciclib in 4 Cohorts of Locoregionally Advanced Inoperable or Metastatic Androgen Receptor-positive Triple-negative Breast Cancer
Brief Title: Bicalutamide and Abemaciclib in Inoperable or Metastatic Androgen Receptor-positive Triple-negative Breast Cancer
Acronym: ABBICAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Kom Op Tegen Kanker (Other); Eli Lilly and Company (Industry); Teva Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S66466; 2022-502272-23-00 (Other: EU CT Number)
Record Dates: First submitted 2023-07-11; First posted 2024-04-15 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-12

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: Triple Negative Breast Cancer; Receptors, Androgen
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Bulbo-Spinal Atrophy, X-Linked | interventions — abemaciclib; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Abemaciclib and bicalutamide (Experimental): Participants receive Abemaciclib 150 mg tablet orally twice daily and Bicalutamide 150 mg orally once daily until disease progression or unacceptable toxicity.
  Interventions: Drug: Abemaciclib; Drug: Bicalutamide

INTERVENTIONS:
Drug: Abemaciclib — 150 mg tablet orally twice daily
  Other Names: Verzenios
Drug: Bicalutamide — 150 mg tablet orally once daily
  Other Names: Bicalutamide Teva

SUMMARY:
This study has as goal to evaluate the use of abemaciclib and bicalutamide in androgen receptor positive metastatic triple negative breast cancer.

DETAILED DESCRIPTION:
This study is a phase II single arm clinical trial. Phase II clinical trials test the safety and effectiveness of an intervention to learn whether the intervention works in treating a specific disease.

In this study, the investigators will include patients with locally advanced unresectable or metastatic androgen receptor positive triple negative breast cancer. The participants need to be progressive after at least 1 prior cytostatic regimen in advanced setting.

The participants will be treated with bicalutamide and abemaciclib. Bicalutamide works against the androgen receptor and abemaciclib stops the cell cycle.

The investigators will look into if this combination can help patients with androgen receptor positive triple negative breast cancer. The investigators will also look into if this is a safe combination.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analysis. If a patient declines to participate in any voluntary exploratory research of the study, there will be no loss of benefit to the patient and she will not be excluded from other aspects of the study
2. Women aged at least 18 years
3. The patient has a biopsy-confirmed diagnosis of recurrent, unresectable, locally advanced, or metastatic AR+ TNBC

   1. AR+ assessed locally and defined as ≥1% of cells staining on IHC of last recurrent/metastatic breast cancer specimen
   2. Local biopsy confirmation of last recurrent/metastatic site with positive IHC for ER and/or PR in ≤10% of cells and negative for HER2 per ASCO/CAP-guidelines
   3. Prior invasive (metastatic) breast cancer with positive IHC for ER and/or PR in >10% of cells is allowed, provided the last biopsy of recurrent/metastatic disease has positive IHC for ER and/or PR in ≤10% of cells
   4. Prior invasive (metastatic) HER2-positive breast cancer per ASCO/CAP-guidelines is not allowed
   5. The patient has measurable disease per RECIST 1.1 or evaluable bone-only disease with lytic or mixed component that is progressive as evidenced on pre-treatment baseline imaging
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks
5. The patient must have had prior treatment with at least 1 prior cytostatic regimen in advanced setting setting unless treatment with a cytostatic regimen is contraindicated as judged by Investigator. There is no upper limit for prior treatment lines in advanced setting.

   * Patients with 1-10% cells with positive IHC for ER in the last recurrent/metastatic site must be treated with at least one line of endocrine therapy in advanced setting.
   * Patients with known germline BRCA1/2 pathogenic variants should have received previous treatment with PARP inhibitors in the early/locally advanced or metastatic setting, unless contraindicated.
   * Prior treatment with palbociclib or ribociclib is allowed, provided at least 6 months have elapsed between last administration and start of study treatment
6. Patients must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of prior anticancer treatment except for residual Grade 2 alopecia, anemia or peripheral neuropathy prior to randomization. A washout period of at least 21 days is required between last chemotherapy dose and first dose of study drug (provided the patient did not receive radiotherapy).
7. Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization.
8. In females of child-bearing potential, a negative serum or urine pregnancy test within 7 days prior to starting treatment is required. Women of child-bearing potential must agree to use a highly effective method of contraception prior to study entry, for the duration of study participation (in addition to the LHRH-agonist), and for 3 weeks following completion of abemaciclib and for 130 days following completion of bicalutamide.

A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

1. Treatment with any of the following:

   a. Any experimental treatment in a clinical trial within the last 30 days or 5 half-lives, whichever is longer, prior to randomization.

   b) Currently enrolled in any other type of medical research (for example: medical device) judged by the sponsor not to be scientifically or medically compatible with this study.

   c. Any other chemotherapy, immunotherapy or anticancer agents within 21 days of the first dose of study treatment d. Treatment with palbociclib or ribociclib within 6 months of the first dose of study treatment e. Any prior exposure to abemaciclib f. Any prior exposure to anti-androgen therapy (bicalutamide, abiraterone, and/or enzalutamide)
2. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment
3. Spinal cord compression, leptomeningeal carcinomatosis, or brain metastases - unless asymptomatic, treated, stable at baseline imaging and not requiring corticosteroids >10 mg prednisolone daily (or equivalent) for at least 2 weeks prior to start of study treatment
4. Concurrent use of endocrine therapy (tamoxifen, anastrozole, letrozole, exemestane, oral contraceptive pills)
5. The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
6. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
7. Any of the following cardiac criteria:

   1. Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 consecutive electrocardiograms (ECGs)
   2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (eg, complete left bundle branch block, third degree heart block)
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval
   4. Personal history of syncope of cardiovascular etiology, ventricular arrhythmia (of pathologic origin including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
   5. Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure NYHA Grade 2 or greater
   6. Uncontrolled hypotension - Systolic BP <90mmHg and/or diastolic BP <50mmHg
   7. Known left ventricular ejection fraction (LVEF) below lower limit of normal for site
8. Prior history of DVT/PE or embolic stroke, unless currently on therapeutic anticoagulation
9. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   1. Absolute neutrophil count < 1.5 x 109/L
   2. Platelet count < 100 x 109/L
   3. Hemoglobin < 8 g/dL (Patients may receive transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.)
   4. Alanine aminotransferase > 3 times the upper limit of normal (ULN)
   5. Aspartate aminotransferase > 3 times ULN
   6. Total bilirubin > 1.5 times ULN (patients with Gilbert's syndrome with a total bilirubin ≤2.0 times ULN and direct bilirubin within normal limits are permitted)
   7. Creatinine >1.5 times ULN concurrent with creatinine clearance < 50 ml/min (measured or calculated per local institutional practice); confirmation of creatinine clearance is only required when creatinine is > 1.5 times ULN
   8. Known proteinuria 3+ on dipstick analysis or >500mg/24 hours
   9. Sodium or potassium outside normal reference range for site. Grade 1 abnormality of sodium and potassium (as defined by CTCAE v5.0) can be included if judged clinically not significant by the investigator, based on the participant's clinical context and comorbidities.
10. Liver disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis. Patients who are hepatitis B Core antibody IgG positive are allowed to participate if taking and compliant with daily oral hepatitis B prophylactic medications
11. Severely impaired lung function defined as spirometry and DLCO that is less than or equal to 50% of the normal predicted value and/or 02 saturation that is 89% or less at rest on room air and/or serious /uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy).
12. Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
13. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of abemaciclib and/or bicalutamide
14. Patients with an active bleeding diathesis
15. The patient has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
16. History of hypersensitivity or allergic reaction to abemacliclib, bicalutamide or goserelin, or drugs with a similar chemical structure or class
17. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
18. Co-administration with strong CYP3A4 inducers (e.g., phenytoin, rifampin, carbamazepine, St John's Wort, bosentan, efavirenz, etravirine, modafinil, and nafcillin) or strong CYP3A4 inhibitors (e.g., clarithromycin, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, verapamil, and voriconazole). See Appendix 4 for complete list.
19. Other invasive malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
20. Female patients who are pregnant or breast feeding/lactating, or females of reproductive potential who are not using effective birth control methods. Hormonal contraceptives are not acceptable as a method of contraception.
21. Patients with hereditary problems of galactose intolerance, total lactase deficiency, or glucose-galactose malabsorption

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with disease control at 16 weeks | Week 16
  Disease control rate at week 16 in all patients (cohorts A, B, C and D combined) treated at the selected dose level. DCR is defined as the proportion of patients that present with stable disease, partial response or complete response per RECIST 1.1 at 16 weeks after treatment initiation.

SECONDARY OUTCOMES:
Number of participants with (serious) adverse events, death and clinical abnormalities per Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | 2 years
  Based on clinically relevant changes from baseline for vital signs and laboratory findings. CTCAE v5.0 uses a range of grades from 1 to 5: grade 1 = mild; grade 2 = moderate; grade 3 = severe; grade 4 = life-threatening; grade 5 = death
HRQoL change from baseline as measured by EORTC QLQ-C30 | 2 years
  The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaires Core-30 item (QLQ-C30) is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  The possible scores for question 1 to 28 are: 1 = not at all; 2 = a little; 3 = quite a bit; 4 = very much. A lower score means a worse outcome.
  The possible scores for question 29 and 30 are between 1 and 7 with 1 = very poor and 7 = excellent. A higher score means a better outcome.
Number of participants with disease control at 16 weeks in subgroup with androgen receptor (AR) positivity on immunohistochemistry (IHC) in ≥10% of cells. | Week 16
  Disease control rate (DCR) at 16 weeks for treatment with abemaciclib in combination with bicalutamide in the subgroup with positive AR IHC in ≥10% of cells. DCR is defined as the proportion of patients that present with stable disease, partial response or complete response per RECIST 1.1 at 16 weeks after treatment initiation.
Number of participants with disease control at 16 weeks in subgroups A, B, C and D separate | Week 16
  Disease control rate (DCR) at 16 weeks for treatment with abemaciclib in combination with bicalutamide in subgroups A, B, C and D separate. DCR is defined as the proportion of patients that present with stable disease, partial response or complete response per RECIST 1.1 at 16 weeks after treatment initiation.
Number of participants with disease control at 24 weeks | Week 16
  Disease control rate (DCR) at 24 weeks for treatment with abemaciclib in combination with bicalutamide in all patients, in the 4 cohorts separate and in the subgroups with IHC for AR ≥10%. DCR is defined as the proportion of patients that present with stable disease, partial response or complete response per RECIST 1.1 at 24 weeks after treatment initiation.
Number of participants with partial or complete response at 16 weeks | Week 16
  Overall response rate (ORR) at 16 weeks in all patients with measurable disease, in the 4 cohorts separate and in the subgroups with IHC for AR ≥10%. ORR is defined as the proportion of patients that present with partial response or complete response per RECIST 1.1 at 16 weeks after treatment initiation.
Duration of response | 2 years
  Duration of response (DOR) in all patients with measurable disease and partial or complete response, in the 4 cohorts separate and in the subgroups with IHC for AR ≥10%. DOR is defined as the time from response until disease progression or death in patients who achieve complete or partial response.
Months of progression free survival | 2 years
  Progression free survival (PFS) in all patients, in the 4 cohorts separate and in the subgroups with IHC for AR ≥10%. PFS is defined as the time from start of treatment until disease progression/relapse or death from any cause. If the specific event (disease progression/relapse, death, whatever comes first) does not occur, PFS will be censored at the date of last tumor assessment. In case no tumor assessment is available, patients will conservatively be censored at the date of first bicalutamide + abemaciclib dose.
Months of overall survival | 2 years
  Overall survival (OS) in all patients, in the 4 cohorts separate and in the subgroups with IHC for AR ≥10%. OS is defined as the time from start of treatment until death from any cause. Patients who are still alive at the time of OS analysis will be censored at the last date they were known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Neven, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (6):
- Belgium (6):
  - ZAS Augustinus, Antwerp
  - Antwerp University Hospital, Antwerp
  - University Hospital Brussels, Brussels
  - Ghent University Hospital, Ghent
  - Jessa Ziekenhuis, Hasselt
  - University Hospitals Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No